CLINICAL TRIAL: NCT03853473
Title: Prehabilitation of Frail Surgical Cancer Patients Using Remote Ischemic Preconditioning
Acronym: Prehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Matthew J. Durand, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO00032510; 1R21AG062933 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Colon Cancer; Fragility; Prehabilitation; Surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Blinded, Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are randomized by the study statistician to receive either the intervention (remote ischemic conditioning) or standard of care. Participants cannot be blinded using this model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Study participants will receive standard of care.
- Remote Ischemic Preconditioning (Experimental): Study participants will perform remote ischemic preconditioning daily, at home, from study enrollment to their date of surgery.
  Interventions: Procedure: Remote Ischemic Preconditioning

INTERVENTIONS:
Procedure: Remote Ischemic Preconditioning — Remote Ischemic Preconditioning (RIPC) occurs when a limb is made transiently ischemic (5 minutes) using a simple blood pressure cuff. We are proposing that study participants in the RIPC group perform the intervention daily at home for at least 14 days prior to scheduled surgery. They will inflate a blood pressure cuff on the upper portion of their nondominant arm, inflate it to 225 mmHg for 5 minutes, release the cuff for 5 minutes, and repeat this 5 times (for a total of 45 minutes). A study coordinator will monitor compliance with phone calls and daily log sheets that must be filled out.
  Arms: Remote Ischemic Preconditioning

SUMMARY:
This project will examine the efficacy of a simple, cost-effective, non-invasive intervention, called remote ischemic preconditioning (RIPC), to reduce frailty in pre-surgical, frail, elderly patients with colon cancer. The investigators hypothesize that RIPC will reduce frailty in the pre-surgical period (as assessed by distance walked during the 6-minute walk test), improve functional capacity 4-weeks postoperatively, and reduce intraoperative blood pressure variability. If successful, future studies will examine the efficacy of RIPC to improve surgical outcomes in frail cancer patients.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) was first described three decades ago as an intervention to protect vital organs from ischemic injury. RIPC occurs when a tissue is made transiently ischemic (5 minutes) for repeated bouts (5 times) prior to the longer ischemic insult. Recently it has been shown exercise performance and motor function are improved in young, healthy individuals when RIPC is performed on the arm or leg using a simple blood pressure cuff to occlude blood flow to the limb. The application of RIPC to individuals with reduced functional capacity, however, is largely unexplored. The study team was the first to apply RIPC to chronic stroke survivors with reduced physical function, and two weeks of RIPC increases walking speed, paretic muscle strength and fatigue resistance. Advanced age and cancer are both dramatic accelerators of frailty and frail patients have poor surgical outcomes. Therefore, the investigators propose to apply this non-invasive, simple intervention as a "prehabilitation" therapy to elderly patients with colon cancer during the perioperative period. The investigators will enroll 96 colon cancer patients aged 55-85 who are ≥17 days prior to scheduled curative resection of colon cancer. After study enrollment, all participants will perform the six-minute walk test as a measure of frailty. Participants will then be randomized to receive either RIPC on their upper, non-dominant arm daily for 14 days prior to surgery, or to receive standard of care (no intervention). After 14 days of either RIPC or no intervention, the 6-minute walk test will be re-assessed within 48 hours of surgery. The primary study outcome will be the difference in six-minute walk distance (in meters) between patients in the RIPC group vs. those in the standard of care group following the two-week pre-operative intervention period (Aim 1). The investigators hypothesize that patients in the RIPC group will walk further during the six-minute walk test than those in the standard of care group due to the well-defined effects of RIPC to improve athletic performance, cardiovascular function, and strength in healthy individuals. A secondary study outcome will be the difference in six-minute walk test distance between the RIPC and standard of care group 4-weeks postoperatively (Aim 2). The investigators hypothesize that patients in the RIPC group will have more rapid recovery from surgery, which would be evidenced by increased walking endurance post-operatively. Another secondary study outcome will be the amount of intraoperative blood pressure variability (time systolic pressure is above or below 135 mmHg or 95 mmHg, respectively) between the RIPC and control groups (Aim 3). The investigators hypothesize that RIPC will reduce intraoperative blood pressure variability due to the well described effects of RIPC to improve systemic vascular function. Future larger studies will examine the effects of RIPC prehabilitation on surgical outcomes such as length of hospital stay and all-cause mortality in frail, elderly patients with colon cancer as well as other patient cohorts with reduced functional capacity.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 55-85
* Have a positive diagnosis of colon cancer or suspected colon cancer based on pathology report
* Be scheduled for curative resection of non-metastatic colon cancer
* Have a 6-Minute Walk Test distance ≤80% of predicted value based on age and sex.

Exclusion Criteria:

* Condition which prevents walking
* Any condition in which compression of the arm or transient ischemia is contraindicated (e.g. wounds in the arm)
* Neurodegenerative disorder
* Unstable angina in previous month
* Myocardial infarction during previous month.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Durand, Ph.D., Principal Investigator — Medical College of Wisconsin; Julie K Freed, MD, Ph.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were consented following their clinical appointments. Group assignment did not occur until after pre-testing, which often occurred on a separate day.
Period: Overall Study
Arm/Group | Standard of Care | Remote Ischemic Preconditioning
Started (Study participants were assigned to either group after they completed baseline testing. Five individuals were consented following their surgical consultation and their baseline testing session was scheduled for a later date due to the timing of their planned surgery. Those participants reconsidered study participation and withdrew. These five individuals account for the discrepancy between total patients enrolled (17) and total patients who started and were assigned to a group (12).) | 6 | 6
Completed | 5 | 4
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Remote Ischemic Preconditioning | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (5) | 71 (8) | 74 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Test Distance (Pre Surgery)
Description: The investigators will compare the distance study participants can walk in 6 minutes in the pre-surgical period as a measure of frailty.
Time Frame: Pre-Surgery
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Standard of Care | Remote Ischemic Preconditioning
Number analyzed (Participants) | 5 | 4
Meters | 369 (60) | 432 (42)

2. Secondary Outcome: 10 Meter Walk Test (Pre Surgery)
Description: The investigators will compare the speed study participants walk over 10 meters in the pre-surgical period as a secondary measure of frailty.
Time Frame: Pre-Surgery
Measure: Mean (Standard Deviation); unit: Meters/Second
Arm/Group | Standard of Care | Remote Ischemic Preconditioning
Number analyzed (Participants) | 5 | 4
Meters/Second | 1.12 (0.17) | 1.27 (0.04)

3. Secondary Outcome: Timed Up and Go (Pre Surgery)
Description: The investigators will compare the speed study participants stand from a chair, walk three meters, turn around, walk back to the chair, and sit (timed up and go test) in the pre-surgical period as a secondary measure of frailty.
Time Frame: Years 1-3
Reporting Status: Not Posted

4. Secondary Outcome: Hand Grip Strength (Pre Surgery)
Description: The investigators will compare handgrip strength in the presurgical period as a secondary measure of frailty.
Time Frame: Years 1-3
Reporting Status: Not Posted

5. Secondary Outcome: 6 Minute Walk Test Distance (Post Surgery)
Description: The investigators will compare the distance study participants walk in 6-minutes 4-weeks post-surgery as a secondary outcome of surgical recovery.
Time Frame: Years 1-3
Reporting Status: Not Posted

6. Secondary Outcome: 10 Meter Walk Test (Post Surgery)
Description: The investigators will compare the speed study participants walk 10 meters 4-weeks post-surgery as a secondary outcome of surgical recovery.
Time Frame: Years 1-3
Reporting Status: Not Posted

7. Secondary Outcome: Timed Up and Go (Post Surgery)
Description: The investigators will compare the speed study participants stand from a chair, walk three meters, turn around, walk back to the chair, and sit (timed up and go test) 4-weeks post surgery as a secondary measure of surgical recovery.
Time Frame: Years 1-3
Reporting Status: Not Posted

8. Secondary Outcome: Hand Grip Strength (Post Surgery)
Description: The investigators will compare handgrip strength 4-weeks post surgery as a secondary measure of surgical recovery.
Time Frame: Years 1-3
Reporting Status: Not Posted

9. Secondary Outcome: Intraoperative Blood Pressure Variability
Description: The investigators will measure the variability of blood pressure during the intraoperative period using the anesthetic record.
Time Frame: Years 1-3
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Number of Hours of Rehabilitation
Description: The investigators will document the number of hours of physical therapy each study participant participates in following surgery.
Time Frame: Years 1-3
Reporting Status: Not Posted

11. Other Pre Specified Outcome: All Cause Mortality
Description: The investigators will document any deaths that occur during hospitalization following surgery.
Time Frame: Years 1-3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Length of Hospital Stay
Description: The investigators will document how long participants in both study groups (RIPC or standard of care) stay in the hospital following surgery.
Time Frame: Years 1-3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from enrollment to study completion, an average of 6-weeks.
Arm/Group | Standard of Care | Remote Ischemic Preconditioning
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=6) | Remote Ischemic Preconditioning (N=6)
Arm turned purple following Ischemic Conditioning (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Participants arm turned purple following IC intervention. Participant was examined by a member of study team who is an MD. Symptoms resolved and participant was withdrawn from study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03853473/Prot_SAP_ICF_000.pdf